CLINICAL TRIAL: NCT01471457
Title: The Use of Trimo-San Gel for the Prevention of Pessary-associated Bacterial Vaginosis
Brief Title: Trial of Trimosan Gel Effect on Pessary-associated Bacterial Vaginosis
Acronym: TBVAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-028
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial; vaginosis; pessary; discharge
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimo-San group (Experimental): Pessary wearers are instructed to apply one fingertip (approx 1 tablespoon) of Trimo-San gel inside the vagina or to the pessary (for women removing and cleaning pessary before reinsertion after cleaning) once nightly
  Interventions: Drug: Trimo-San gel
- Control group (No Intervention): Pessary wearers are informed on standard care of pessary, which includes topical estrogen application if they are using. Pessary wearers do not use Trimo-San gel

INTERVENTIONS:
Drug: Trimo-San gel — Pessary wearers are instructed to apply one fingertip (approx 1 tablespoon) of Trimo-San gel inside the vagina or to the pessary (for women removing and cleaning pessary before reinsertion after cleaning) once nightly
  Arms: Trimo-San group

SUMMARY:
The primary objective of this prospective, randomized, controlled study is to assess the effect of Trimo-San vaginal gel on the rate of bacterial vaginosis in women who use pessaries. Women being fitted for a pessary for the first time or not wearing a pessary for >1 year are recruited in to the study and randomized to using Trimo-San gel daily or not using Trimo-San gel. The investigators use two objective measures of bacterial vaginosis (OSOM BV blue and gram stain) and subjective questionnaires regarding the presence and effect of vaginal symptoms on the pessary user prior to pessary fitting and at 3 months post pessary fitting. The investigators hypothesize that Trimo-San gel with not significantly affect the rate of bacterial vaginosis in pessary wearers as measures by OSOM BV blue and Gram stain, but will have a positive effect on the subjective symptoms experienced by women wearing pessaries.

DETAILED DESCRIPTION:
The study population will consist of women who will be fitted for and initiate use of a pessary for relief of pelvic organ prolapse and/or urinary symptoms.

All patients scheduled for pessary fitting/initiation who meet the above inclusion criteria will be asked to participate in the study. They are randomized using opaque envelopes pulled sequentially, which were made originally from a blocked design, stratified to women removing the pessary daily themselves and women not removing the pessary daily themselves. Prior to pessary fitting all women in the study answer a brief questionnaire about their vaginal symptoms. Subjects undergo a vaginal swab for OSOM BV Blue (copyright by Genzyme, SekiSui) and Gram stain testing for Nugent's criteria the presence of bacterial vaginosis. Women are then fitted with and instructed on use of a pessary in the standard fashion by a trained physician at at the study sites.

Women will be randomized to either standard pessary care or to use of TrimoSan gel twice a week (half applicator) to the vagina either with applicator or applying half applicator amount to the surface of the pessary before insertion. If women are using additional vaginal medications such as Premarin this information will be collected but not change their randomization and they will continue to use other indicated vaginal medications as they did before participation in the study (per clinical judgement).

At 2 weeks and 3 month after pessary initiation the patients are seen for an office visit. At both the 2 week and 3 month visit they have repeat testing for bacterial vaginosis using vaginal swab for OSOM BV Blue (copyright by Genzyme) and Gram stain testing. At both the 2 week and 3 month visits they will also answer a questionnaire about their vaginal symptoms and the effect of these symptoms on their distress and lifestyle. This questionnaire is similar to the baseline questionnaire answered before initiation of pessary use, and will include questions about whether these symptoms have changed since initiation of their pessary. At the University of New Mexico site, information is also being collected on sexual function using the PISQ-IR questionnaire and on body image using the modified Body Image Scale at baseline, 2 weeks, and 3 months. At this particular site women will also answer questions about their management of the pessary (e.g. if they take it out for intercourse) surrounding sexual activity.

The recruitment goal for this study is 150 women, with 75 in each group. This was calculated to detect a significant difference in the rate of bacterial vaginosis between the control and study groups (α=0.05), and assuming baseline of bacterial vaginosis to be approximately 10% in the population and increased to 30% by hypothetical risk factors, the sample size needed for each group is 62 for a power of 80%. Assuming a 15% dropout rate after recruitment, we plan to randomize at least 75 patients to the control group and 75 patients to the study group for a total of at least 150 patients. 60 women were recruited for this study at the initial site of Washington Hospital Center in Washington, D.C. This study site closed in June 2012. In January 2013 the study opened at University of New Mexico in Albuquerque, NM. The study is currently opening and running at University of New Mexico with the recruitment goal of 90 women at this institution.

The primary outcome measure will be rate of bacterial vaginosis in the study population, to be compared between the control (non Trimo-San using) and study (Trimo-San using) groups. As part of this analysis, we will also compare the rate of bacterial vaginosis in the control and study groups before and after pessary initiation. Secondary outcomes will include:

* Change in vaginal symptoms as assessed by questionnaire before and after initiation of pessary use
* Change in level of worry or distress about vaginal symptoms as assessed by questionnaire before and after initiation of pessary use.
* Change in vaginal symptoms or distress about these symptoms as assessed by questionnaire based on use or non-use of Trimo-San gel.
* Describe the management of women of their pessary surrounding sexual activity (University of New Mexico only)
* Change in body image or sexual function associated with initiation of the pessary or use of TrimoSan gel (University of New Mexico only)

ELIGIBILITY:
Inclusion Criteria:

* Female
* Indications for initiation of pessary use and planning to be fitted for and wear a pessary

Exclusion Criteria:

* Male
* Already using a pessary or have used in the last year
* History of recurrent or chronic bacterial vaginosis with > 2 episodes per year or symptoms reported for > 6 months out of last year
* Active known vaginal infection (symptomatic and/or untreated) or completion of treatment for BV or cervical/vaginal infection within one week of recruitment
* History of active vaginal ulcerative disease (active ulcers from atrophy, herpes symptoms at recruitment, or HSV with > 2 outbreaks per year or last outbreak < 1 month ago)
* Chronic antibiotic use for indications not listed above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate V Meriwether, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of New Mexico, Albuquerque, New Mexico

REFERENCES:
- [Background] Alnaif B, Drutz HP. Bacterial vaginosis increases in pessary users. Int Urogynecol J Pelvic Floor Dysfunct. 2000;11(4):219-22; discussion 222-3. doi: 10.1007/pl00004026. PMID 11005473
- [Background] Eschenbach DA, Hillier S, Critchlow C, Stevens C, DeRouen T, Holmes KK. Diagnosis and clinical manifestations of bacterial vaginosis. Am J Obstet Gynecol. 1988 Apr;158(4):819-28. doi: 10.1016/0002-9378(88)90078-6. PMID 3259075
- [Background] Landers DV, Wiesenfeld HC, Heine RP, Krohn MA, Hillier SL. Predictive value of the clinical diagnosis of lower genital tract infection in women. Am J Obstet Gynecol. 2004 Apr;190(4):1004-10. doi: 10.1016/j.ajog.2004.02.015. PMID 15118630
- [Background] Powers K, Lazarou G, Wang A, LaCombe J, Bensinger G, Greston WM, Mikhail MS. Pessary use in advanced pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Feb;17(2):160-4. doi: 10.1007/s00192-005-1311-8. Epub 2005 May 10. PMID 15883856
- [Background] Myziuk L, Romanowski B, Johnson SC. BVBlue test for diagnosis of bacterial vaginosis. J Clin Microbiol. 2003 May;41(5):1925-8. doi: 10.1128/JCM.41.5.1925-1928.2003. PMID 12734228
- [Background] Bradshaw CS, Morton AN, Garland SM, Horvath LB, Kuzevska I, Fairley CK. Evaluation of a point-of-care test, BVBlue, and clinical and laboratory criteria for diagnosis of bacterial vaginosis. J Clin Microbiol. 2005 Mar;43(3):1304-8. doi: 10.1128/JCM.43.3.1304-1308.2005. PMID 15750100
- [Background] Forsum U, Hallen A, Larsson PG. Bacterial vaginosis--a laboratory and clinical diagnostics enigma. APMIS. 2005 Mar;113(3):153-61. doi: 10.1111/j.1600-0463.2005.apm1130301.x. PMID 15799757
- [Derived] Bugge C, Adams EJ, Gopinath D, Stewart F, Dembinsky M, Sobiesuo P, Kearney R. Pessaries (mechanical devices) for managing pelvic organ prolapse in women. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD004010. doi: 10.1002/14651858.CD004010.pub4. PMID 33207004
- [Derived] Gupta A, Cox C, Dunivan GC, Gaskins JT, Rogers RG, Iglesia CB, Meriwether KV. Desire for Continued Pessary Use Among Women of Hispanic and Non-Hispanic Ethnic Backgrounds for Pelvic Floor Disorders. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):172-177. doi: 10.1097/SPV.0000000000000652. PMID 30807423
- [Derived] Fregosi NJ, Hobson DTG, Kinman CL, Gaskins JT, Stewart JR, Meriwether KV. Changes in the Vaginal Microenvironment as Related to Frequency of Pessary Removal. Female Pelvic Med Reconstr Surg. 2018 Mar/Apr;24(2):166-171. doi: 10.1097/SPV.0000000000000520. PMID 29474292
- [Derived] Meriwether KV, Rogers RG, Craig E, Peterson SD, Gutman RE, Iglesia CB. The effect of hydroxyquinoline-based gel on pessary-associated bacterial vaginosis: a multicenter randomized controlled trial. Am J Obstet Gynecol. 2015 Nov;213(5):729.e1-9. doi: 10.1016/j.ajog.2015.04.032. Epub 2015 Apr 30. PMID 25935783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trimo-San Group | Control Group
Started | 92 | 92
Completed | 73 | 74
Not Completed | 19 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trimo-San Group | Control Group | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15) | 60 (17) | 59 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 184
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 56 | 48 | 104
  Black/African American | 6 | 13 | 19
  Hispanic | 23 | 20 | 43
  Asian | 1 | 3 | 4
  Other | 5 | 8 | 13
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meters] | 29 (7.6) | 28 (7.4) | 28 (7.5)
Smoking [Count of Participants; unit: Participants]
  Current smoker | 8 | 6 | 14
  Past Smoker | 26 | 28 | 54
  Non-smoker (never smoker) | 58 | 58 | 116
Charleston Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — Minimum 0; maximum 30 points Higher scores worse, one point assigned for each disease with exception of 2 points for hemiplegia, mod to severe renal disease, diabetes with end organ damage, or any cancer, and 6 points each for metastatic cancer or AIDS
  units on a scale | 0.77 (1.1) | 0.89 (1.8) | 0.82 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Bacterial Vaginosis at 3 Months
Description: The primary outcome is the rate of bacterial vaginosis after pessary fitting as measured by OSOM BV blue (Genzyme) and gram stain, measured in women using and women not using Trimo-San gel after pessary fitting, at 3 months, with the denominator being the number of women having a gram stain at the 3 months time point in each group
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Trimo-San Group | Control Group
Number analyzed (Participants) | 62 | 71
Participants | 15 | 16

2. Secondary Outcome: Participants With Any Bothersome Vaginal Symptom at 3 Months
Description: Vaginal symptoms and effect of vaginal symptoms on pessary wearers measured before and after pessary fitting by questionnaire based on verified vaginal symptoms questionnaire at 3 months, with the denominator being the number of women completing the questionnaire at the 3 months time point in each group
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Trimo-San Group | Control Group
Number analyzed (Participants) | 72 | 75
Participants | 30 | 24

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events are worsening of vaginal symptoms since pessary fitting; this could be treatment related or not treatment related Serious adverse events were any recorded events that required hospitalization or were life-threatening, whether related or unrelated to treatment
Arm/Group | Trimo-San Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 18/92 | 13/92
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trimo-San Group (N=92) | Control Group (N=92)
Any vaginal symptom attributable possibly to pessary (Reproductive system and breast disorders) | 18 (18) | 13 (13) — At least one or more vaginal symtoms (itching, pain, discharge, etc) that has increased since pessary fitting at 9 mo

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No